CLINICAL TRIAL: NCT01663987
Title: A Randomized, Placebo-controlled, Double-blind, Parallel Group, Multi Center Study to Assess the Safety and Efficacy of Tiotropium Bromide (18 µg) Delivered Via the HandiHaler® in Chronic Obstructive Pulmonary Disease (COPD) Subjects Recovering From Hospitalization for an Acute Exacerbation (Hospital Discharge Study 1)
Brief Title: Investigate the Impact of Early Treatment Initiation With Tiotropium in Patients Recovering From Hospitalization for an Acute COPD Exacerbation 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.477
Record Dates: First submitted 2012-08-09; First posted 2012-08-14 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

ARMS (2):
- 18 mcg tiotropium (Active Comparator): Patient to receive one tiotropium bromide inhalation powder capsule daily (in the morning) via HandiHaler
  Interventions: Drug: tiotropium bromide
- Placebo (Placebo Comparator): Patient to receive one placebo capsule daily (in the morning) identical to those containing tiotropium bromide inhalation powder via HandiHaler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tiotropium bromide — 18 mcg once a day (QD)
  Arms: 18 mcg tiotropium
Drug: Placebo — once a day (QD)
  Arms: Placebo

SUMMARY:
A randomized, placebo-controlled, double-blind, parallel group, multi center study to assess the safety and efficacy of tiotropium bromide (18 µg) delivered via the HandiHaler® in Chronic Obstructive Pulmonary Disease (COPD) subjects recovering from hospitalization for an acute exacerbation (Hospital Discharge 1)

ELIGIBILITY:
Inclusion criteria:

The following inclusion criteria apply at Visit 0:

1. All subjects must sign an informed consent consistent with the International Conference on Harmonization - Good Clinical Practice (ICH-GCP) guidelines prior to participation in the trial and conducting any study procedures.
2. Male or female subjects 40 years of age or older.
3. Hospitalization for a primary diagnosis of acute COPD exacerbation for =14 days. Determination of accuracy of admission diagnosis will be at the discretion of the investigator.
4. Patient reported hospital length of stay and discharge date (confirmed with hospital discharge summary/hospital records; however, medical record confirmation may occur following randomization).

   The following inclusion criteria apply at Visit 1:
5. Discharged from the hospital =10 days from date of randomization.
6. All subjects must have a diagnosis of COPD (P12-01205), and have documented airway obstruction with a post-bronchodilator Force expiratory volume in 1 second (FEV1)/Force vital capacity (FVC )<0.7(See Section 5.1.2, Pulmonary Function Testing). The diagnosis of COPD can be made at Visit 1 if no Pulmonary Function Testing (PFT) data available within the past 12 months.
7. Subjects must be current or ex-smoker with a smoking history of =10 pack-years:

Pack-years = Number of cigarettes/day x years of smoking 20 cigarettes/ pack 8. Subjects must be able to inhale medication in a competent manner from the HandiHaler® device (Appendix 10.1) and from a metered dose inhaler (MDI).

Exclusion criteria:

The following exclusion criterion applies at Visit 0:

1. No more than 30 days of therapy with any long-acting inhaled anticholinergic over preceding 3 months prior to discharge from the hospital, and no therapy with any long acting anticholinergic post discharge (no use between hospital discharge and randomization) or any other restricted concomitant medications

   The following exclusion criteria apply at Visit 1:
2. Presence of a significant disease (in the opinion of the investigator) which may put the subject at risk because of participation in the study or may influence the subject's ability to participate in the study for up to 2 years.
3. A documented history of myocardial infarction during the hospitalization preceding randomization. Subjects being stable with a history of cardiac stents are permitted.
4. Any unstable or life-threatening cardiac arrhythmia requiring intervention or change in drug therapy during the last year.
5. Subjects with asthma (subject treated for asthma in the last 2 years, history of childhood asthma is permitted), cystic fibrosis, clinical diagnosis of bronchiectasis, interstitial lung disease, pulmonary thromboembolic disease or known active tuberculosis.

7. Malignancy for which the subject has undergone resection, radiation, chemotherapy or biological treatments within the last two years or is currently on active radiation therapy, chemotherapy or biological treatment. Subjects with treated basal cell carcinoma and non-invasive squamous cell skin carcinoma are allowed.

8. Hospitalization for cardiac failure (New York Heart Association (NYHA) class III or IV) during the hospitalization preceding randomization.

9. Known hypersensitivity to anticholinergic drugs, lactose, or any other components of the HandiHaler® or MDI inhalation solution delivery system.

10. Known moderate to severe renal impairment as judged by the investigator. 11. Known narrow angle glaucoma as judged by the investigator. 12. Significant symptomatic prostatic hyperplasia or bladder-neck obstruction. Subjects whose symptoms are controlled on treatment may be included. 13. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e., oral contraceptives, intrauterine devices, diaphragm or sub dermal implants e.g., Norplant) for at least three months prior to and for the duration of the trial.

14. Significant alcohol or drug abuse within the past 12 months. 15. Previously randomized in this study or currently participating in another interventional study.

16. Visual impairment that as judged by the investigator does not allow the subject to independently read and complete the questionnaires and eDiary.

17. Any significant or new ECG findings at Visit 1 as judged by the investigator, including, but not limited to signs of acute ischemia, arrhythmia.

18. Treatment with any restricted pulmonary medication. 19. Residing in an assisted living facility.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2014-05-01 (Actual); Study Completion 2014-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (50):
- United States (49):
  - 205.477.001039 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 205.477.001050 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 205.477.001021 Boehringer Ingelheim Investigational Site, Florence, Alabama
  - 205.477.001046 Boehringer Ingelheim Investigational Site, Fountain Valley, California
  - 205.477.001052 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 205.477.001059 Boehringer Ingelheim Investigational Site, San Diego, California
  - 205.477.001009 Boehringer Ingelheim Investigational Site, Stamford, Connecticut
  - 205.477.001040 Boehringer Ingelheim Investigational Site, Waterbury, Connecticut
  - 205.477.001051 Boehringer Ingelheim Investigational Site, Brandon, Florida
  - 205.477.001044 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 205.477.001037 Boehringer Ingelheim Investigational Site, Eustis, Florida
  - 205.477.001017 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 205.477.001063 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 205.477.001001 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 205.477.001004 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 205.477.001012 Boehringer Ingelheim Investigational Site, Duluth, Georgia
  - 205.477.001064 Boehringer Ingelheim Investigational Site, Belleville, Illinois
  - 205.477.001038 Boehringer Ingelheim Investigational Site, Muncie, Indiana
  - 205.477.001007 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 205.477.001014 Boehringer Ingelheim Investigational Site, Columbia, Maryland
  - 205.477.001018 Boehringer Ingelheim Investigational Site, Livonia, Michigan
  - 205.477.001068 Boehringer Ingelheim Investigational Site, Union, New Jersey
  - 205.477.001035 Boehringer Ingelheim Investigational Site, Cooperstown, New York
  - 205.477.001023 Boehringer Ingelheim Investigational Site, New York, New York
  - 205.477.001061 Boehringer Ingelheim Investigational Site, Staten Island, New York
  - 205.477.001027 Boehringer Ingelheim Investigational Site, Burlington, North Carolina
  - 205.477.001032 Boehringer Ingelheim Investigational Site, Huntersville, North Carolina
  - 205.477.001020 Boehringer Ingelheim Investigational Site, Seneca, North Carolina
  - 205.477.001034 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 205.477.001053 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 205.477.001011 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 205.477.001057 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 205.477.001006 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 205.477.001083 Boehringer Ingelheim Investigational Site, Downingtown, Pennsylvania
  - 205.477.001031 Boehringer Ingelheim Investigational Site, Monroeville, Pennsylvania
  - 205.477.001028 Boehringer Ingelheim Investigational Site, Anderson, South Carolina
  - 205.477.001019 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 205.477.001010 Boehringer Ingelheim Investigational Site, Fort Mill, South Carolina
  - 205.477.001025 Boehringer Ingelheim Investigational Site, Gaffney, South Carolina
  - 205.477.001002 Boehringer Ingelheim Investigational Site, Rock Hill, South Carolina
  - 205.477.001026 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 205.477.001015 Boehringer Ingelheim Investigational Site, Union, South Carolina
  - 205.477.001013 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 205.477.001022 Boehringer Ingelheim Investigational Site, Corsicana, Texas
  - 205.477.001055 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 205.477.001054 Boehringer Ingelheim Investigational Site, Katy, Texas
  - 205.477.001062 Boehringer Ingelheim Investigational Site, Tyler, Texas
  - 205.477.001030 Boehringer Ingelheim Investigational Site, Abingdon, Virginia
  - 205.477.001008 Boehringer Ingelheim Investigational Site, Roanoke, Virginia
- 205.477.001043 Boehringer Ingelheim Investigational Site, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomized, placebo-controlled, double blind, parallel group design involving an event-driven treatment period up to the close of the study and a minimum 30-day follow-up period up to the close of the study
Groups:
- Placebo: Patient to receive oral inhalation of one placebo powder capsule once daily in the morning via HandiHaler.
- Tiotropium Bromide (18μg): Patient to receive oral inhalation of one tiotropium bromide powder capsule once daily in the morning via HandiHaler.
Period: Overall Study
Arm/Group | Placebo | Tiotropium Bromide (18μg)
Started | 39 | 40
Completed | 26 | 34
Not Completed | 13 | 6
Not completed — Adverse Event | 7 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Other reason not defined above | 3 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The treated set included all patients randomized and who took at least one dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tiotropium Bromide (18μg) | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (7.5) | 58.9 (11.5) | 58.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Trough FEV1 at 12 Weeks on Study Drug
Description: Change from baseline in trough forced expiratory volume in 1 second (FEV1) at 12 weeks on study medication. Trough FEV1 is defined as FEV1 measurement prior to the next dosing of study drug and approximately 24 hours after the last inhalation of drug.
Time Frame: Baseline and 12 weeks
Population: Treated Set (TS) including patients who had trough FEV1 data at both baseline and week 12
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo | Tiotropium Bromide (18μg)
Number analyzed (Participants) | 30 | 30
Litres | -0.051 (0.224) | 0.183 (0.273)

2. Primary Outcome: Percentage of Patients With Next Adverse Clinical Outcome Event From the Two Twin Trials, Present 205.477 (NCT01663987) and 205.478 (NCT01662986)
Description: Percentage of patients with next adverse clinical outcome event occured during the study, defined as the combined endpoint of chronic obstructive pulmonary disease (COPD) exacerbations per Boehringer Ingelheim (BI) definition, all-cause re-hospitalization, or all-cause mortality.
  Time to the next adverse clinical outcome event from the two twin trials, was defined as a primary endpoint but was not analysed numerically, so this endpoint is presented instead.
  This endpoint was analysed using combined data, as specified in the analysis plan.
Time Frame: From first drug administration to the last timepoint with information of clinical adverse outcome available, up to 2 years
Population: Treated set of the pooled twin studies 205.478 and 205.477: This set includes all patients who were randomised and took at least one dose of study drug, 157 patients (79 Tiotropium and 78 placebo) were included in this set.
Measure: Number; unit: Percentage of perticipants
Arm/Group | Placebo | Tiotropium Bromide (18μg)
Number analyzed (Participants) | 78 | 79
Percentage of perticipants | 47.4 | 53.2

3. Secondary Outcome: Change From Baseline of Trough FVC at 12 Weeks on Study Drug
Description: Change from baseline of trough Forced Vital Capacity (FVC) at 12 weeks on study drug.
Time Frame: Baseline and 12 weeks
Population: Treated Set (TS) including patients who had trough FVC data at both baseline and week 12
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo | Tiotropium Bromide (18μg)
Number analyzed (Participants) | 30 | 30
Litres | -0.117 (0.371) | 0.274 (0.308)

4. Secondary Outcome: Percentage of Patients With Adverse Clinical Event on Study
Description: Percentage of patients with adverse clinical event during on study, which is defined as the combined endpoint of chronic obstructive pulmonary disease (COPD) exacerbations per Boehringer Ingelheim (BI) definition, all-cause re-hospitalisation, or all cause mortality.
Time Frame: as for outcome 2
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tiotropium Bromide (18μg)
Number analyzed (Participants) | 39 | 40
Percentage of participants | 59.0 | 60.0

5. Secondary Outcome: Change From Baseline of Trough FEV1 at 12 Weeks on Study Drug From the Two Twin Trials, Present 205.477 (NCT01663987) and 205.478 (NCT01662986)
Description: Change from baseline of Trough FEV1 (forced expiratory volume in one second) at 12 weeks on study drug.
  Trough FEV1 is defined as the FEV1 measurement prior to the next dosing of study drug and approximately 24 hours after last inhalation of drug.
  This endpoint was analysed using combined data, as specified in the analysis plan.
Time Frame: Baseline and 12 weeks
Population: Treated Set of the pooled twin studies 205.478 and 205.477. The number of patients analyzed at week 12 from the treated set were 59 for Placebo and 60 for Tiotropium.
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo | Tiotropium Bromide (18μg)
Number analyzed (Participants) | 59 | 60
Litres | 0.035 (0.262) | 0.185 (0.384)

6. Secondary Outcome: Change From Baseline of Trough FVC at 12 Weeks From the Two Twin Trials, Present 205.477 (NCT01663987) and 205.478 (NCT01662986)
Description: Change from baseline of trough Forced Vital Capacity (FVC) at 12 weeks on study drug.
  This endpoint was analysed using combined data, as specified in the analysis plan.
Time Frame: Baseline and 12 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo | Tiotropium Bromide (18μg)
Number analyzed (Participants) | 59 | 60
Litres | -0.015 (0.396) | 0.278 (0.447)

7. Secondary Outcome: Percentage of Patients With COPD Exacerbation From the Two Twin Trials, Present 205.477 (NCT01663987) and 205.478 (NCT01662986)
Description: Percentage of patients with COPD exacerbation on study was analysed for the combined study.
  A COPD exacerbation was defined as a complex of lower respiratory events/symptoms (increase or new onset) related to the underlying COPD with duration of three days or more, requiring a change in treatment where a complex of lower respiratory events/symptoms was defined as at least two of the following: 1) Shortness of breath; 2) Sputum production (volume); 3)Occurrence of purulent sputum; 4) Cough; 5) Wheezing; 6) Chest tightness. Onset of exacerbation was defined by the onset of first recorded symptom.The end of exacerbation was decided by the investigator based on clinical judgment.
  A required change in treatment included either prescription of antibiotics and/or systemic steroids; and a newly prescribed maintenance respiratory medication (i.e. bronchodilators including theophyllines and PDE4-inhibitors).
  This endpoint was analysed using combined data, as specified in the analysis plan.
Time Frame: as for outcome 2
Population: Treated set of the pooled twin studies 205.478 and 205.477
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tiotropium Bromide (18μg)
Number analyzed (Participants) | 78 | 79
Percentage of participants | 44.9 | 40.5

8. Secondary Outcome: Percentage of Patients With All-cause Hospitalization From the Two Twin Trials, Present 205.477 (NCT01663987) and 205.478 (NCT01662986)
Description: Percentage of patients with all-cause hospitalization outcome event occured during the study was analysed for the combined study.
  All-cause hospitalization included all hospitalizations, except planned hospitalizations for elective procedures. Hospitalizations occurring on the same day as discharge were not considered a separate admission.
  This endpoint was analysed using combined data, as specified in the analysis plan.
Time Frame: as for outcome 2
Population: Treated set of the pooled twin studies 205.478 and 205.477
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tiotropium Bromide (18μg)
Number analyzed (Participants) | 78 | 79
Percentage of participants | 26.9 | 26.6

9. Secondary Outcome: Percentage of Patients With 30-day Readmission Rates Outcome Event From the Two Twin Trials, Present 205.477 (NCT01663987) and 205.478 (NCT01662986)
Description: Percentage of patients with 30-day hospital readmission rates outcome events was analysed.
  Days to hospital readmission were calculated as:Hospital readmission days = Readmission date - Date of hospital discharge + 1.
  The 30-day hospital readmission analysis summarized the frequency of patients with hospital readmission and readmission days >1 and <31 days using the TS.
  This endpoint was analysed using combined data, as specified in the analysis plan.
Time Frame: from date of hospital discharge prior to randomization up to readmission days >1 and <31 days
Population: Treated set of the pooled twin studies 205.478 and 205.477
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tiotropium Bromide (18μg)
Number analyzed (Participants) | 78 | 79
Percentage of participants | 5.1 | 5.1

10. Secondary Outcome: Number of COPD Exacerbation Events From the Two Twin Trials, Present 205.477 (NCT01663987) and 205.478 (NCT01662986)
Description: Number of COPD exacerbation per patient year outcome event occured during the study was analysed descriptively by calculating average occurrence (number of events per patient year drug exposure) by treatment group for on study period using the TS.
  This endpoint was analysed using combined data, as specified in the analysis plan.
Time Frame: Start of treatment to the last timepoint with information of clinical adverse outcome available, up to 2 years
Population: Treated Set of the pooled twin studies 205.478 and 205.477. The number of patients analyzed for this endpoint from the treated set were 73 for Placebo and 54 for Tiotropium.
Measure: Number; unit: exacerbations per patient year
Arm/Group | Placebo | Tiotropium Bromide (18μg)
Number analyzed (Participants) | 73 | 54
exacerbations per patient year | 1.3 | 0.9

11. Secondary Outcome: Number of All-cause Hospitalization Event From the Two Twin Trials, Present 205.477 (NCT01663987) and 205.478 (NCT01662986)
Description: Number of all-cause hospitalization per patient year outcome event occured during the study was analysed descriptively by calculating average occurrence (number of events per patient year drug exposure) by treatment group for on study period using the TS.
  This endpoint was analysed using combined data, as specified in the analysis plan.
Time Frame: as for outcome 2
Population: Treated Set of the pooled twin studies 205.478 and 205.477. The number of patients analyzed for this endpoint from the treated set were 47 for Placebo and 38 for Tiotropium.
Measure: Number; unit: Hospitalisation per patient year
Arm/Group | Placebo | Tiotropium Bromide (18μg)
Number analyzed (Participants) | 47 | 38
Hospitalisation per patient year | 0.8 | 0.6

12. Secondary Outcome: Time to Event: Time to Recovery (EXACT-PRO) From the Two Twin Trials, Present 205.477 (NCT01663987) and 205.478 (NCT01662986)
Description: Time to event: Time to recovery based on EXACT-PRO total score. The percentage of observed patients recovered by end of study was reported.
  Time to recovery was assessed with the EXACT-PRO questionnaire. EXACT-PRO total scores were transformed to smooth scores for determining time to recovery and all other endpoints related to the EXACT questionnaire. The day-2 score was transformed to the mean of the total scores recorded on Day 1, 2, and 3. Similarly, each subsequent day's score was transformed to the mean score using a rolling 3-day average.
  Analysis based on Kaplan Meier estimate.
Time Frame: From first drug administration to the last timepoint with information of EXACT-PRO, up to 2 years
Population: This endpoint was not analysed due to the trials being terminated prematurely due to low patient enrollment and the limited amount of data.
Measure: Number; unit: Percentage of patients recovered
Arm/Group | Placebo | Tiotropium Bromide (18μg)
Number analyzed (Participants) | 76 | 76
Percentage of patients recovered | 94.0 | 88.0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after the last dose of study drug, up to 524 days
Arm/Group | Placebo | Tiotropium Bromide (18μg)
Serious Adverse Events (participants affected / at risk) | 15/39 | 15/40
Other Adverse Events (participants affected / at risk) | 21/39 | 19/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=39) | Tiotropium Bromide (18μg) (N=40)
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 2 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Incision site infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 11 | 12
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=39) | Tiotropium Bromide (18μg) (N=40)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2
Bronchitis (Infections and infestations) | 2 | 3
Candida infection (Infections and infestations) | 3 | 1
Oral candidiasis (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 2 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 17 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
The original protocol planned to randomize 604 subjects, however this was not reached due to low patient enrollment. All results are descriptive only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.